CLINICAL TRIAL: NCT03237624
Title: Use of a Functional Chewing Gum in Reduction of Gingival Inflammation
Brief Title: Functional Chewing Gum in Reduction of Gingival Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Harlan Shiau, Clinical Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HP-00073354
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Gingivitis
Keywords: gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional chewing gum (Experimental): Subjects given as intervention functional chewing gum device to supplement oral hygiene practices. Functional gum contains chitosan which is a food additive or generally recognized as safe food product. Individuals will use this gum 20 to 30 minutes three times per day. Subjects will brush and floss normally twice a day.
  Interventions: Device: Functional Chitosan Chewing Gum; Behavioral: Oral hygiene measures
- Control chewing gum (Placebo Comparator): Subjects given control gum to supplement oral hygiene practices. Placebo gum does not contain any active ingredients. Individuals will use this gum 20 to 30 minutes three times per day. Subjects will brush and floss normally twice a day.
  Interventions: Device: Control Chewing Gum; Behavioral: Oral hygiene measures

INTERVENTIONS:
Device: Functional Chitosan Chewing Gum — Chitosan and chitosan-related preparations have been shown to have some antimicrobial properties, possibly in the disruption of bacterial colonization. It is thought that as a component of a functional chewing gum this will supplement in the removal of daily build up of dental plaque on tooth surfaces.
  Arms: Functional chewing gum
Device: Control Chewing Gum — Control chewing gum device does not have food additive chitosan in its composition.
  Arms: Control chewing gum
Behavioral: Oral hygiene measures — Patients will be given instructions on how to brush and floss routinely (twice per day)

SUMMARY:
The aim of this prospective randomized 3-month double-blinded single center study is to determine whether a chewing gum device with food additive chitosan, will aid in reducing gingival inflammation by supplementing traditional tooth brushing and flossing measures. Patients with mild to moderate gingivitis will be identified and enrolled in this investigation. All enrolled subjects will receive baseline oral hygiene brushing instructions and a baseline clinical examination of the gingiva. The test group will utilize the test chewing gum three times a day for a minimum 20-30 minutes duration; the control group will receive a placebo gum and use it in a similar manner. We will examine whether daily use of a functional chewing gum enhances improvements to brushing and flossing.

DETAILED DESCRIPTION:
Periodontal disease remains a prevalent and preventable disease in man. Plaque bacterial biofilm remains the primary etiologic agent of disease; colonization of non-shedding tooth surfaces greatly contributes to initiation and progression of gingivitis, for example. Although there are currently available chemotherapeutic agents to supplement daily oral hygiene measures, one continuous issue is patient compliance. Chewing gum represents a unique delivery device for not only drugs and other agents, but food additives that might aid in reducing bacteria plaque colonization on tooth surfaces. For example, chitosan and chitosan-related food additive preparations have been shown to have some antimicrobial-like properties, possibly in the disruption of bacterial colonization (not -cidal).

NOTE: ALL INGREDIENTS of the "test" chewing gum, and the placebo chewing gum, are generally regarded as safe ("GRAS" label by the Food and Drug Administration), as they are common food components. For example, chitosan is listed in the GRAS database (https://www.accessdata.fda.gov/scripts/fdcc/?set=SCOGS). See item GRN No. 397.

This study aims to determine whether adjunctive use of functional chewing gum will improve gingival inflammation status-retaining clinical gains initiated by professional tooth cleaning and at home brushing over a 12 week period in gingivitis patients.

Eligibility criteria and outcome measures are described in the next section.

ELIGIBILITY:
Inclusion Criteria:

* Mild-moderate gingivitis
* Minimum of 20 natural teeth

Exclusion Criteria:

* Significant alveolar bone loss as evidenced by Bite-wings (>3.0 mm cementoenamel junction to bone)
* Requirement for antibiotic pre-medication prior to dental procedures
* Systemic antibiotic use in past 14 days to current.
* Use of oral contraceptives
* Use of anti-inflammatory (NSAIDs) or in past 14 days.
* Use of anticoagulant therapy or in past 14 days.
* Poorly controlled diabetes (HbA1c > 7.9%)*
* Smoking
* Pregnancy
* Use of any oral rinses such as, but not limited to chlorhexidine, essential oils, cetylpyridinium chloride during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Gum inflammation change | Change in color of gingiva from baseline to 12 weeks
  Measure the color of gingiva - use Gingiva Index

SECONDARY OUTCOMES:
Plaque levels (on teeth) change | Change in plaque level from baseline to 12 weeks
  Measure plaque using Plaque Index

CONTACTS AND LOCATIONS:
Overall Officials: Harlan Shiau, DDS, Principal Investigator — UMSOD
Locations (1):
- University of Maryland School of Dentistry, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaur S, Dhillon GS. The versatile biopolymer chitosan: potential sources, evaluation of extraction methods and applications. Crit Rev Microbiol. 2014 May;40(2):155-75. doi: 10.3109/1040841X.2013.770385. Epub 2013 Mar 14. PMID 23488873
- [Background] Machul A, Mikolajczyk D, Regiel-Futyra A, Heczko PB, Strus M, Arruebo M, Stochel G, Kyziol A. Study on inhibitory activity of chitosan-based materials against biofilm producing Pseudomonas aeruginosa strains. J Biomater Appl. 2015 Sep;30(3):269-78. doi: 10.1177/0885328215578781. Epub 2015 Apr 8. PMID 25855683
- [Background] Li Y, Lee S, Hujoel P, Su M, Zhang W, Kim J, Zhang YP, DeVizio W. Prevalence and severity of gingivitis in American adults. Am J Dent. 2010 Feb;23(1):9-13. PMID 20437720
- [Background] Simons D, Beighton D, Kidd EA, Collier FI. The effect of xylitol and chlorhexidine acetate/xylitol chewing gums on plaque accumulation and gingival inflammation. J Clin Periodontol. 1999 Jun;26(6):388-91. doi: 10.1034/j.1600-051x.1999.260609.x. PMID 10382579